CLINICAL TRIAL: NCT02315144
Title: A 2-Stage, Single-Dose Study in Healthy Volunteers and COPD Patients With an Open Label Ipratropium Bromide Reference to Evaluate the Efficacy, Pharmacokinetics, and Safety Profile of Inhaled TV48108
Brief Title: An Efficacy and Safety Profile of Inhaled TV48108 in Healthy Volunteers and COPD Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TV48108-COPD-10045
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; bronchodilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- TV48108 - Healthy Volunteers (Experimental): Stage 1 is a randomized, placebo-controlled, double-blind, single-dose study. Healthy subjects will be randomized to receive a single inhaled dose of TV48108 120 µg
  Interventions: Drug: TV48108
- Placebo - Healthy Volunteers (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- TV48108 15 µg COPD (Experimental): Stage 2 consists of a 2-period open-label study with an ipratropium bromide reference to evaluate the single administration of 3 ascending doses of inhaled TV48108 in COPD patients.
  Interventions: Drug: TV48108
- TV48108 60 µg COPD (Experimental): Stage 2
  Interventions: Drug: TV48108
- TV48108 120 µg COPD (Experimental): Stage 2 .
  Interventions: Drug: TV48108

INTERVENTIONS:
Drug: TV48108 — TV48108 15, 60, 120 μg
  Other Names: 48108
  Arms: TV48108 - Healthy Volunteers; TV48108 120 µg COPD; TV48108 15 µg COPD; TV48108 60 µg COPD
Drug: Placebo — Placebo Comparator
  Other Names: Matching placebo
  Arms: Placebo - Healthy Volunteers

SUMMARY:
The primary objective of the study is to characterize the safety profile and duration of bronchodilation of a single dose of inhaled TV48108.

ELIGIBILITY:
Inclusion Criteria:

Stage 1 (Healthy Volunteers)

* Male or female 20 to 75 years of age, inclusive, weighing 50 to 80 kg with a body mass index (BMI) of less than 30 kg/m^2.
* In good health as determined by medical and psychiatric history, physical examination, electrocardiogram (ECG), serum chemistry, hematology, urinalysis, and serology.
* Other criteria apply, please contact the investigator for more information

Stage 2 (Chronic Obstructive Lung Disease (COPD) patients)

* Male or female; 40 to 75 years of age, inclusive with a minimum body weight of 40 kg
* Current or former cigarette smokers with a history of cigarette smoking of ≥10 pack years at the screening visit
* Diagnosis of COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease guidelines.
* Other criteria apply, please contact the investigator for more information

Exclusion Criteria:

Stage 1 (Healthy Volunteers)

* History or current evidence of a clinically significant or uncontrolled disease
* Any disorder that may interfere with the absorption, distribution, metabolism or excretion of study drugs.
* History of severe allergy to milk protein
* Active smokers or former smokers who quit within 3 months of the first dose of study drug. Former smokers with greater than five-pack years (ie, the equivalent of one pack per day for five years) are also excluded.
* Other criteria apply, please contact the investigator for more information

Stage 2 (Chronic Obstructive Lung Disease (COPD) patients)

* Recent history of hospitalization due to an exacerbation of airway disease within 3 months
* Need for increased treatments of COPD within 6 weeks prior to the screening visit
* History of and/or current diagnosis of asthma
* Known α1 antitrypsin deficiency, active lung infections (such as tuberculosis or pneumonia), and lung cancer are absolute exclusionary conditions
* Other criteria apply, please contact the investigator for more information

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Baseline adjusted forced expiratory volume in 1 second area under the curve over 12 hours (FEV1 AUC0-12h). | Day 1 (pre-dose, up to 12 hours post-dose)

SECONDARY OUTCOMES:
Baseline Adjusted Trough 12 hour forced expiratory volume in 1 second (FEV1) | Day 1 (pre-dose, up to 12 hours post-dose)
Percentage of Participants with Adverse Events | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (7):
- United States (2):
  - Teva Investigational Site 13038, Medford, Oregon
  - Teva Investigational Site 13039, Spartanburg, South Carolina
- Australia (3):
  - Teva Investigational Site 78992, Clayton
  - Teva Investigational Site 78993, Daws Park
  - Teva Investigational Site 78991, Melbourne
- New Zealand (2):
  - Teva Investigational Site 79041, Auckland
  - Teva Investigational Site 79040, Christchurch